CLINICAL TRIAL: NCT03819959
Title: Metabolomics Pilot Study on Intensive Care Acquired Muscle Weakness in Polytrauma (MIRACLE-II Study)
Brief Title: Metabolomics Study on Intensive Care Acquired Muscle Weakness in Polytrauma
Acronym: MIRACLE II
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, Stefan Schaller, Principal Investigator, Technical University of Munich
Other Study IDs: MIRACLE II
Record Dates: First submitted 2019-01-19; First posted 2019-01-29 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Metabolomics; Critical Care; Critical Illness; Critical Illness Myopathy; Critical Illness Polyneuropathy; Intensive Care (ICU) Myopathy; Muscle Weakness
Keywords: Pilot Trial; Muscle Biopsy; Blood Metabolome
MeSH Terms: conditions — Critical Illness; Polyneuropathies; Muscular Diseases; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood
  * Skeletal muscle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive Care Patients: Polytrauma patients who have been admitted to intensive care

SUMMARY:
In this mono-center pilot trial, polytrauma patients admitted to intensive care will be included. Investigators are going to take blood and muscle samples at respecified time points to do metabolic, histological and molecular testing.

Aim of the study is to investigate (1) changes of the blood metabolome in patients with ICUAW (intensive care unit acquired weakness) and (2) identify metabolic components who are responsible for ICUAW or can be used as marker for ICUAW.

ELIGIBILITY:
Inclusion Criteria:

* acute polytrauma patient
* age ≥ 18 years old
* expected intensive care stay ≥ 3 days
* American Society of Anesthesiologists classification I or II

Exclusion Criteria:

* patient had received cardiopulmonary resuscitation
* limitation of therapy or comfort care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: polytrauma patients who are admitted to intensive care
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Metabolomics | a median of 14 days
  Blood Metabolome will be isolated from blood samples. All samples will be screened for changes in the blood metabolome during muscle wasting (i.e. Intensive Care Unit Acquired Weakness) using mass spectrometry

SECONDARY OUTCOMES:
Muscle histology | a median of 14 days
  Immunohistochemistry will be done in muscle samples. All samples will be screened for changes in the muscular structure and correlation with blood metabolome changes.
Phosphoproteomics | a median of 14 days
  Phosphoproteomics will be done in muscle samples using mass spectrometry. All samples will be screened for influence of muscular changes (i.e. Intensive Care Unit Acquired Weakness (ICUAW)) and correlation with blood metabolome changes.

OTHER OUTCOMES:
Identify possible predictors of muscle wasting in the blood metabolome at ICU admission | a median of 14 days
  Identify metabolites or combinations of metabolites whose high or low concentration(s) at ICU admission associate(s) with the amount of muscle loss. These metabolites are candidate biomarkers that could be used to identify individuals at risk of large muscle wasting and may give further insights into the mechanisms of muscle wasting.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, MHBA, Principal Investigator — Technical University of Munich; Hennig Wackerhage, PhD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, School of Medicine, Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided